CLINICAL TRIAL: NCT07077421
Title: Investigation of the Relationship Between Postoperative Pain and Both Central Sensitization Severity and Sleep Quality in Patients Undergoing Breast Cancer Surgery
Brief Title: Postoperative Pain, Central Sensitization, and Sleep Quality in Breast Cancer Surgery Patients
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nur Hilal Durukan Gündoğan, Medical Doctor, Istanbul University - Cerrahpasa
Other Study IDs: 2025/81
Record Dates: First submitted 2025-06-28; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Pain; Breast Cancer Surgery; Central Sensitization; Sleep Quality
MeSH Terms: conditions — Pain, Postoperative; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Good Sleep Quality Group: Participants with Pittsburgh Sleep Quality Index (PSQI) score less than 5, indicating good sleep quality. No intervention is applied to alter sleep patterns; this is a stratification based on preoperative sleep assessment.
- Poor Sleep Quality Group: Participants with PSQI score of 5 or greater, indicating poor sleep quality. This group is used to assess the relationship between preoperative sleep disturbance and postoperative pain outcomes. No intervention is applied.
- Low Central Sensitization Severity Group: Participants with Central Sensitization Inventory (CSI) score below 40, indicating low central sensitization severity. Used for comparative analysis of postoperative pain scores. No therapeutic intervention applied.
- High Central Sensitization Severity Group: Participants with CSI score of 40 or greater, indicating high central sensitization severity This grouping aims to evaluate the effect of central sensitization on postoperative pain perception and analgesic needs. No intervention administered.

SUMMARY:
This prospective observational study aims to investigate whether preoperative central sensitization and sleep quality are associated with acute postoperative pain levels in patients undergoing breast cancer surgery.

The study includes 41 female patients scheduled for unilateral breast cancer surgery. Before surgery, participants are evaluated using two self-report questionnaires: the Central Sensitization Inventory (CSI) and the Pittsburgh Sleep Quality Index (PSQI). Based on their scores, participants are categorized into groups according to central sensitization level and sleep quality.

After surgery, all participants receive a standardized multimodal analgesia protocol. Pain severity is measured using the Numeric Rating Scale (NRS) at five time points within the first 24 hours: 30 minutes, 2, 6, 12, and 24 hours postoperatively. Additional assessments include sedation level (Ramsay Sedation Scale), nausea and vomiting (Verbal Descriptive Scale), and presence of delirium (Nursing Delirium Screening Scale - NuDESC).

The primary question this study seeks to answer is whether higher levels of central sensitization and/or poor sleep quality prior to surgery are predictive of greater acute postoperative pain.

DETAILED DESCRIPTION:
This prospective observational cohort study is designed to evaluate the association between preoperative central sensitization levels, sleep quality, and acute postoperative pain intensity in female patients undergoing breast cancer surgery. The study is being conducted at Istanbul University-Cerrahpaşa, Cerrahpaşa Medical Faculty, Department of Anesthesiology and Reanimation, in collaboration with the Department of General Surgery, from March 2025 to June 2025, following ethics committee approval and prospective registration.

A total of 41 female patients, aged between 18 and 80 years, undergoing unilateral breast surgery with sentinel lymph node biopsy (SLNB)-including simple mastectomy, breast-conserving surgery, or mastectomy with immediate reconstruction-are included. All participants provide written informed consent before enrollment.

Preoperative assessments are performed one day prior to surgery. Central sensitization is measured using the Central Sensitization Inventory (CSI), a 25-item self-report questionnaire assessing symptoms commonly associated with central sensitization. A CSI-A score ≥40 is considered indicative of high central sensitization. Sleep quality is evaluated with the Pittsburgh Sleep Quality Index (PSQI), a validated instrument assessing sleep characteristics over the past month; PSQI scores ≥5 are accepted as reflecting poor sleep quality.

All patients receive standardized general anesthesia and multimodal analgesia including:

Induction: Fentanyl 2 mcg/kg (lean body weight), propofol 2 mg/kg (lean body weight), rocuronium 0.6 mg/kg (actual body weight).

Maintenance: Sevoflurane and additional opioid supplementation as needed. Intraoperative analgesia: Morphine 0.05 mg/kg (lean body weight). Postoperative analgesia: Scheduled paracetamol and NSAIDs; opioids as rescue medication if required.

Pain severity is measured using the Numeric Rating Scale (NRS) at five postoperative time points: 30 minutes, 2, 6, 12, and 24 hours. Additional assessments include:

Sedation level: Ramsay Sedation Scale (RSS) Nausea and vomiting: Verbal Descriptive Scale (VDS) Delirium screening: Nursing Delirium Screening Scale (NuDESC) Participants are categorized into groups according to their CSI and PSQI scores. Postoperative pain scores and secondary outcomes are compared across these groups using non-parametric statistical methods (e.g., Mann-Whitney U test for independent samples). Correlation analyses (Spearman's rank) are performed to assess relationships between CSI, PSQI, and postoperative pain scores.

The primary objective is to determine whether high central sensitization and/or poor sleep quality are predictive of increased acute postoperative pain. Secondary objectives include evaluating the relationship between preoperative risk factors and sedation, nausea/vomiting, and delirium outcomes.

A power analysis was conducted based on expected effect sizes from previous literature, targeting a minimum of 31 participants for 80% statistical power with an alpha of 0.05. A 20% dropout margin was included, resulting in a final sample size of 41 participants.

All data are collected using standardized case report forms. Data entry is conducted by trained personnel and monitored for consistency and completeness. Ethical approval was obtained from the institutional review board prior to participant recruitment. The study does not receive external funding.

ELIGIBILITY:
InclusionCriteria:

* Female patients aged between 18 and 80 years
* Scheduled to undergo one of the following unilateral breast cancer surgeries with sentinel lymph node biopsy (SLNB):
* Simple mastectomy
* Breast-conserving surgery (BCS)
* Simple mastectomy with immediate breast reconstruction
* ASA Physical Status Classification I-III
* Able to understand the study procedure and provide informed consent
* Fluent in Turkish and capable of completing self-report questionnaires
* Preoperative completion of the following assessments:
* Central Sensitization Inventory (CSI)
* Pittsburgh Sleep Quality Index (PSQI)

ExclusionCriteria:

* Pregnant or lactating women
* Allergy or contraindication to any component of the analgesic regimen (e.g., paracetamol, dexketoprofen, tramadol, fentanyl, or morphine)
* Planned or performed intraoperative regional nerve block (e.g., paravertebral or PECS block)
* Use of sedative-hypnotic drugs, opioids, or gabapentinoids within the last 7 days
* History of prior breast or axillary surgery
* Conversion to emergency surgery or development of major intraoperative complications
* Admission to the intensive care unit (ICU) postoperatively
* Patient refusal to participate in postoperative assessments
* Evidence of metastatic disease

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of female patients aged 18 to 80 years who were admitted for elective breast cancer surgery at the Department of Anesthesiology and Reanimation, Istanbul University-Cerrahpaşa, Cerrahpaşa Medical Faculty Hospital. Participants were selected consecutively among those scheduled for unilateral simple mastectomy, breast-conserving surgery, or mastectomy combined with immediate breast reconstruction. All surgeries were performed under general anesthesia. Preoperative evaluations and postoperative follow-up (within 24 hours) were conducted in a tertiary-care academic hospital setting. Patients were evaluated using standardized self-report questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2025-03-13 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Postoperative Acute Pain Intensity Measured by the Numeric Rating Scale (NRS) | Day 0 (30 minutes, 2 hours, 6 hours, 12 hours, and 24 hours post-surgery)
  Postoperative acute pain intensity will be assessed using the Numeric Rating Scale (NRS; range 0-10, where 0 = no pain and 10 = worst imaginable pain) at rest and during movement. Measurements will be taken at 30 minutes, 2 hours, 6 hours, 12 hours, and 24 hours after surgery.

SECONDARY OUTCOMES:
Sedation Level Assessed by Ramsay Sedation Scale (RSS) | Day 0 (30 minutes, 2 hours, 6 hours, 12 hours, and 24 hours post-surgery
  Sedation level will be assessed using the Ramsay Sedation Scale (RSS; range 1-6, where higher scores indicate deeper levels of sedation). Assessments will be conducted at 30 minutes, 2 hours, 6 hours, 12 hours, and 24 hours after surgery.
Postoperative Nausea and Vomiting Severity Scored on a 4-Point Scale (0-3) | Day 0 (30 minutes, 2 hours, 6 hours, 12 hours, and 24 hours post-surgery)
  Postoperative nausea and vomiting (PONV) will be assessed using a 4-point verbal rating scale. Patients will be asked to rate their overall PONV severity as follows:
  0 = No nausea or vomiting
  1. = Mild nausea only, no vomiting
  2. = Moderate nausea and/or one episode of vomiting
  3. = Severe nausea and/or two or more episodes of vomiting
  Higher scores indicate more severe PONV. Evaluations will be performed at 30 minutes, 2 hours, 6 hours, 12 hours, and 24 hours after surgery.
Delirium Assessment Using the Nursing Delirium Screening Scale (NuDESC) | Day 0 (30 minutes, 2 hours, 6 hours, 12 hours, and 24 hours post-surgery)
  Delirium will be assessed using the Nursing Delirium Screening Scale (NuDESC), a validated 5-item observational tool. Each item is scored from 0 to 2, yielding a total score range of 0-10. A total score ≥2 is considered indicative of delirium. Assessments will be conducted at 30 minutes, 2 hours, 6 hours, 12 hours, and 24 hours after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Üniversitesi-Cerrahpaşa Cerrahpaşa Tıp Fakültesi, Istanbul, Turkey (Türkiye)